CLINICAL TRIAL: NCT01577017
Title: Study On The Effects of Letrozole And Clomiphene Citrate For Induction of Ovulation In Polycystic Ovarian Syndrome(PCOS)
Brief Title: The Effects of Letrozole And Clomiphene Citrate For Induction of Ovulation In Polycystic Ovarian Syndrome(PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nik Hazlina (Other)
Responsible Party: Sponsor-Investigator, Nik Hazlina, Associate Professor Dr, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCOS- Letrozole vs Clomid
Record Dates: First submitted 2012-04-04; First posted 2012-04-13 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: ovulation induction, clomiphene citrate, letrozole
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Letrozole (Experimental): Group L will be assigned with Letrozole 5 mg on night on day 5 to day 9 of the cycle
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Women in group L will be assigned with Letrozole on night at day 5 to day 9 of the cycle
  Other Names: Femara (Aromatase Inhibitor)

SUMMARY:
As both medications i.e. CC and letrozole have been shown to be effective in inducing ovulation in PCOS patients, this study was performed in order to evaluate which regime (whether CC or letrozole) is the best to be used as the first line treatment for PCOS patients with infertility for local population. The best regime will therefore could be included in the protocol of management of infertility patients with PCOS so that the quality of patients' care could be improved.

DETAILED DESCRIPTION:
Polycystic Ovarian Syndrome (PCOS) is the most common endocrinopathy among women of reproductive age group and is one of the leading causes of infertility. It is characterized by chronic anovulation and hyperandrogenism with variable clinical manifestations that include oligomenorrhea, infertility, hirsutism, and acne (Ehrmann DA 2005).

Several methods have been described to induce ovulation in PCOS patients- weight reduction, laparoscopic ovarian drilling and the use of various induction ovulation agents like clomiphene citrate (CC), aromatase inhibitors (AIs) and gonadotrophins.

Clomiphene citrate (CC) has been most widely used and standard drug for the treatment of infertility. It is known that clomiphene citrate results in an ovulation rate of 60-85%, but a conception rate of only around 20% (Bayar et al 2006, Sohrabvand et al 2006). About 20-25% of women are resistant to CC and do not ovulate. Discrepancy between ovulation and pregnancy rate is related to anti-estrogenic activity on endometrium and cervical mucus is due to CC has a long half life of 5 to 7 days.

In view of disappointing result of CC treatment with many adverse effect and cost and possible complication of gonadotrophin, the concept of aromatase inhibition was proposed as a new method of ovulation that are easy to use, less expensive and more effective drugs.

Letrozole is an oral, potent, reversible, and highly selective aromatase inhobitor that prevent androgen-to-estrogen (E) conversion. These aromatase inhibitors have a short half life (45 hours), hence is rapidly eliminated from the body. No adverse effect on E target tissues is seen with letrozole due to this short half life; furthermore, it does not down regulate the ER compare to CC.

The main impetus for the development of aromatase inhibitor as ovulation induction agents was to avoid the peripheral antiestrogenic effects of CC, especially the frequent occurrence of a thin endometrial lining (Sohrabvand et al 2006).

Rationale of performing the study As both medications i.e. CC and letrozole have been shown to be effective in inducing ovulation in PCOS patients, this study was performed in order to evaluate which regime (whether CC or letrozole) is the best to be used as the first line treatment for PCOS patients with infertility for local population. The best regime will therefore could be included in the protocol of management of infertility patients with PCOS so that the quality of patients' care could be improved.

HYPOTHESIS

Letrozole is more effective than clomiphene citrate as ovulation agent in PCOS patients.

General Objective To compare the effectiveness of letrozole and clomiphene citrate as ovulation agent in PCOS.

Specific Objectives

i. To identify the ovulation percentage between letrozole and CC ii. To compare the endometrial thickness between letrozole and CC iii. To determine the pregnancy outcome between letrozole and CC iv. To study the associated factors that can affect the effectiveness of the treatment e.g. age, body weight, smoking, duration of marriage, duration of infertility and types of infertility either primary or secondary)

Methodology

1.0 Study design

Prospective, multicenter, randomized control trial.

2.0 Population and sample

Reference population

The reference population will be the female patient diagnosed to have polycystic ovarian syndrome at infertility clinic HSB, Kedah and infertility clinic HUSM, Kelantan and infertility Clinic, Hospital Tengku Ampuan Afzan (HTAA), Kuantan, Pahang.

3.0 Selection criteria 3.1 Inclusion criteria i. Age > 18 years but < 40 years old ii. Was diagnosed PCOS iii. Patient is not illiterate. iv. Normal husband's seminal fluid analysis (SFA) - (Count > 20 million/ml, Motility > 40% and normal morphology > 30%) 3.2 Exclusion criteria : i. Having medical problem eg- renal disease, tyhroid disorder, hyperprolactinemia, liver disease.

ii. Other causes of anovulatory infertility

4.0 Sampling and Sample size

4.1 Sample size

Sample size calculation:

1. Ovulation percentage

   From Hananel Holzer 2006

   Proportion of ovulation rate by using Clomiphene citrate (Po) = 0.60 Proportion of ovualtion rate by using Letrozole (P1) = 0.84

   P = P1 + Po = 0.83 + 0.64 = 0.72 zα = 1.96 zβ = 0.84 for 80% power 2 2 Significance level (α) = 5% (0.05) Power of study ( 1 - β )= 80% β =20% ( 0.2 ) n = (zα√2P(1-P) + zβ√P1(1-P1)+Po(1-Po))2 (P1-Po)2 n = ( 1.96√2(0.72)(1-0.72) + 0.84√0.83(1-0.84) + 0.60(1-0.60))2 (0.75 - 0.50 )2 n = 54 Therefore sample size = 108 + 20 % drop out = 130 By using PS software - sample size : 130
2. Endomterial thickness between letrozole and CC From Mosammat Rhasid et al 2008 Letrozole 2.5 mg, mean ± SD ratio -10.37 ± 1.2 CC 100mg, mean ± SD ratio - 9.03 ± 0.89

   * - 0.5 n = 2 α2 (zα + zβ)2
   * 2 = 2 (1.2)2 ( 1.96 + 0.84) 2 (0.5)2 = 49 per group Therefore sample size = 98 + 20 % drop out Total n = 117 By using software, n = 51 per group, total n = 122
3. Pregnancy rate between letrozole and CC From Mosammat Rashida Begum 2008 Letrozole 2.5mg - pregnancy rate - 40.6% CC 100mg - pregnancy rate - 18.7% ( Po ) = 0.18 (P1) = 0.41 P = P1 + Po = 0.41 + 0.18 = 0.30 zα = 1.96 zβ = 0.84 for 80% power 2 2 Significance level (α) = 5% (0.05) Power of study ( 1 - β )= 80% β =20% ( 0.2 ) n = (zα√2P(1-P) + zβ√P1(1-P1)+Po(1-Po))2 (P1-Po)2 n = ( 1.96√2(0.30)(1-0.30) + 0.84√0.41(1-0.41) + 0.18(1-0.18))2 (0.41-0.18 )2 n = 61 Therefore sample size = 120 + 20 % drop out n= 146

   * The maximun sample size that were calculated for this study is 146. Therefore sample size that were decided for the the study = 150 patients

4.2 Sampling frame All PCOS patients attending Infertility Clinic Hospital Sultanah Bahiyah (HSB), Kedah, Infertility Clinic Hospital Universiti Sains Malaysia (HUSM), Kelantan and Infertility Clinic Hospital Tengku Ampuan Afzan (HTAA), Kuantan, Pahang who fulfill inclusion and exclusion criteria will be recruited in the study.

5.0 Methods of data collection

The study will be conducted after the approval from Hospital Sultanah Bahiyah, Kedah, USM and HTAA, Pahang ethical committee.

All PCOS patients, age more than 18 years old at Gynecology Clinic, HUSM were given information form regarding the study conducted. When the participants agree to involve in this study, the consent form will be given to them. Participants are required to fill the social demographic data which includes age, address, occupation, monthly family income, education status, and duration of marriage, number of parity and year of last child birth. Measurement such as waist circumference, weight, height and blood pressure reading will be recorded. Then patients will be randomized into two groups

Randomization PCOS women who are eligible and fulfilling the criteria of the study will recruit. After they had given inform consent, they will assigned to one of the groups of sealed opaque envelope labelled as C and L. Women in group C will assigned CC 100mg and those in L assigned Letrozole 2.5 mg. The randomization will be done by computer- generated randomization using http://www.randomization.com according to the random sequence.

Group 1- Letrozole group

* The patients will be given letrozole 2.5 mg from D5-D9 of menses.
* Base line TVS at D2 will be done, following spontaneous menses/induction with MPA 10 mg Daily for 1 week.
* Transvaginal scan was done to document the evidence of ovulation only if patient having menses (D8 -10 onwards ).
* If dominant follicle (DF) present (DF> 12mm), repeat TVS every 2 days,
* ovulation is diagnosed when the mature DF is about 18 to 22 mm and then evidence of ruptured about 3 to 4 days later

  o If dominant follicle (DF) absent (DF<12mm), repeat TVS every 3-4 days later.
* Measure Endometrial thickness (ET) for every follow-up.
* If absent of Dominant follicle (DF<12mm up to Days 20), consider failed or anovulation.

Group 2 Clomiphene Citrate Group

* The patients will be given CC 100 mg from D5-D9 of menses.
* Base line TVS at D2 will be done, following spontaneous menses /induction with MPA 10 mg Daily for 1 week.
* Transvaginal scan was done to document the evidence of ovulation only if patient having menses (D8 -10 onwards).
* If dominant follicle (DF) present (DF> 12mm), repeat TVS every 2 days,
* ovulation is diagnosed when the mature DF is about 18 to 22 mm and then evidence of ruptured about 3 to 4 days later
* If dominant follicle (DF) absent (DF<12mm), repeat TVS every 3-4 days later.
* Measure Endometrial thickness (ET) for every follow-up.
* If absent of dominant follicle (DF<12mm up to Days 20), consider failed or anovulation.

In all groups a urine pregnancy test was done 3 weeks after documented ovulation and the patient remained amenorrheic. All study medications will be discontinued when there was a positive pregnancy test. Pregnant patients were then will be followed up until an ultrasound could document the viability of pregnancy. Copies of patients' obstetric records, including delivery records, were reviewed by the investigators to obtain obstetrics outcomes e.g: miscarriage, ectopic pregnancy, molar pregnancy, preterm delivery etc).

Research tool

* General Questionnaire
* Weighing scale using Seca weighing machine
* Measuring tape
* Ultrasound machine
* BP set Investigations Urine pregnancy test Hormonal and biochemical profiles

ELIGIBILITY:
Inclusion criteria

* Age > 18 years but < 40 years old
* Was diagnosed PCOS
* Normal husband's seminal fluid analysis (SFA)

Exclusion criteria :

* Not having medical problems eg- renal disease, tyhroid disorder, hyperprolactinemia, liver disease.
* Other causes of anovulatory infertility

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of ovulation induction among PCOS patients | 6 weeks
  To evaluate the effectiveness of letrozole and clomiphene citrate for induction of ovulation in PCOS patients.

SECONDARY OUTCOMES:
Number of patients that can ovulate and pregnant | 6 weeks
  i. ovulation rate among PCOS patients with letrozole and CC ii. endometrial thickness among patients with letrozole and CC iii. number of pregnancy between letrozole and CC iv. associated factors that can influence the effectiveness of the treatment found in age, body weight, duration of marriage, duration of infertility and types of infertility either primary or secondary among PCOS patients.